CLINICAL TRIAL: NCT04850313
Title: A Prospective, Randomized, Controlled Clinical Study to Evaluate the Use of ProKera Plus® in the Management of Bacterial Corneal Ulcers
Brief Title: Evaluating the Use of ProKera Plus® in the Management of Bacterial Corneal Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study terminated due to slow enrollment
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 262292
Record Dates: First submitted 2021-04-07; First posted 2021-04-20 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-03

CONDITIONS: Bacterial Corneal Ulcer

STUDY DESIGN:
Intervention Model Description: Phase 1: This phase will establish baseline characteristics for each patient that is randomized into the treatment arm for the phase 2 part of the study.
  Phase 2: This phase will test the intervention of using ProKera Plus® versus continuing conventional treatment for the corneal ulcer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Treatment (No Intervention): * Corneal ulcer scraping sent for microbial culture
  * Admission to the hospital for initiation of fortified vancomycin 25mg/mL every 1 hour alternating with fortified tobramycin 15mg/mL every 1 hour, preservative free artificial tears every 2 hours, and doxycycline 100mg twice daily.
  After 48 hours of conventional treatment, consent will be obtained regarding the use of experimental treatment with ProKera Plus® versus continuing conventional method of treatment
- ProKera Plus® Treatment (Experimental): 1. Experimental Treatment Arm , ProKera Plus® will be placed in the eye with the corneal ulcer
  Interventions: Device: ProProKera Plus®

INTERVENTIONS:
Device: ProProKera Plus® — ProKera® is a sutureless form of CryoTek amniotic membrane that is clipped into a dual polycarbonate ring system with the epithelial side up when in contact with the ocular surface.
  Other Names: ProKera Plus®
  Arms: ProKera Plus® Treatment

SUMMARY:
The study design is a prospective, randomized, controlled interventional study to compare the outcome of ProKera Plus® with conventional treatment in patients with vision-threatening bacterial corneal ulcers. The study will be conducted at the University of Arkansas Medical Sciences (UAMS) in two phases for patients who present to an Ophthalmology clinic or Emergency Department at UAMS.

DETAILED DESCRIPTION:
Bacterial keratitis is a serious bacterial infection of the cornea, usually caused by a persistent epithelial defect or ulcer that can lead to permanent vision loss from corneal scarring, perforation or endophthalmitis. An infectious corneal ulcer requires immediate treatment with intensive topical fortified broad-spectrum antibiotics to try to eliminate the pathogen. Corneal tissue destruction can be caused directly by infectious agents, the associated inflammatory response, or by ocular toxicity from frequent dosing of fortified antibiotics.1 Sutured amniotic membrane transplantation (AMT) has been shown to reduce pain and promote healing in human bacterial keratitis.2 ProKera® is a sutureless form of CryoTek amniotic membrane that is clipped into a dual polycarbonate ring system with the epithelial side up when in contact with the ocular surface. ProKera Plus® contains a double layer of CryoTek amniotic membrane tissue to provide extra therapeutic benefit. ProKera Plus® has several advantages over sutured AMT including ease of administration in a clinic setting and reduced overall procedural cost.

The role of ProKera® in the treatment algorithm of corneal ulcers has yet to be fully clarified. There are currently no prospective case studies comparing the use of ProKera® to standard of care conventional treatments in corneal ulcers. The utility of this device would provide valuable information in the treatment of bacterial corneal ulcers.

The objectives are:

1. To determine if ProKera Plus® can lead to better visual recovery when used with bacterial corneal ulcers compared to conventional treatment
2. To determine if ProKera Plus® can actively modify corneal wound healing during the course of managing bacterial corneal ulcers and decrease the overall time to re-epithelialization
3. To determine if ProKera Plus® can decrease pain associated with bacterial corneal ulcers compared to conventional treatment
4. To determine if ProKera Plus® can decrease the amount of corneal opacity and corneal thinning associated with bacterial corneal ulcers compared to conventional treatment
5. To determine if ProKera Plus® can decrease the need for further interventions or surgeries related to complications from bacterial corneal ulcers

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  * Subjects 18 years of age or older, all sexes and races
  * Willing to sign a written informed consent to participate
  * Corneal ulcer criteria: at least 3mm in diameter, opacification located within 3mm of visual axis, infiltrate occupying at least 50% of the corneal thickness, moderate AC cell reaction, clinical picture consistent with bacterial infection later confirmed by culture and gram stain.

Exclusion Criteria:

* History of Immunodeficiency
* History of connective tissue disorders or severe atopic disease
* History of chemical eye injuries
* History of known limbal stem cell deficiency
* History of neurotrophic keratopathy
* History of recent eye surgery, or glaucoma surgery with bleb or drainage tube
* Risk factors and clinical appearance consistent with fungal keratitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Warrner, MD, Principal Investigator — University Of Arkansas For Medical Sciences, Jones Eye Institute
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total number of candidates screened and enrolled in study was 3. The goal of the study was to enroll 24 subjects, 12 subjects per group. Patients were recruited in the medical clinic (UAMS). recruitment started in November 2021 and ended in March 2022.
Pre-assignment Details: After at least 48 hours of conventional treatment, consent will be obtained regarding the use of experimental treatment with Prokera Plus versus continuing conventional treatment. This will be randomized in a 1:1 ratio by a block-randomization schedule to assign subjects to each of the two treatment groups. All three subjects that were screened were consented and assigned a group.
Period: Overall Study
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Started | 1 | 2
Completed | 1 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Treatment | ProKera Plus® Treatment | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Vision Acuity at Baseline [Mean (Standard Deviation); unit: LogMAR] — Visual acuity (VA) was assessed for participants applicable study eye using a Snellen letter chart. VA was collected in Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity.
  LogMAR | 1.9 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 1.45 (.45) | 1.6 (.424)

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity - Visit 1
Description: Visual acuity (VA) was assessed for participants applicable study eye using a Snellen letter chart. VA was collected in Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity.
Time Frame: 5-day Follow-Up, plus or minus 3 days
Population: All randomized subjects regardless of actual treatment, with data at the 5-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
LogMar | 1.3 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 3.3 (.65)

2. Primary Outcome: Visual Recovery - Visit 2
Description: as for outcome 1
Time Frame: 16-day follow-up plus or minus 5 days
Population: All randomized subjects regardless of actual treatment, with data at the 16-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
LogMar | 1.3 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 2.1 (0.2)

3. Primary Outcome: Visual Recovery - Visit 3
Description: as for outcome 1
Time Frame: 30-day follow-up plus or minus 7 days
Population: All randomized subjects regardless of actual treatment, with data at the 30-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
LogMar | 0.6 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 2.1 (0.2)

4. Primary Outcome: Visual Recovery - Visit 4
Description: as for outcome 1
Time Frame: 90 day follow-up plus or minus 10 days
Population: All randomized subjects regardless of actual treatment, with data at the 90-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 1
LogMar | .47 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | .70 (NA) — Standard deviation not available because only one participant was seen due to adverse event and was seen in clinic as part of standard of care only (Not study related).

5. Primary Outcome: Visual Recovery - Visit 5
Description: as for outcome 1
Time Frame: 180-day follow-up plus or minus 14 days
Population: All randomized subjects regardless of actual treatment, with data at the 180-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: LogMar
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 1
LogMar | .6 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 1 (NA) — Standard deviation not available because only one participant was seen due to adverse event and was seen in clinic as part of standard of care only (Not study related).

6. Secondary Outcome: Corneal Re-epithelialization - Visit 1
Description: number of participants who had slit lamp photography which measured fluorescein staining size.
Time Frame: 5-day follow-up plus or minus 3 days
Measure: Number; unit: participants
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
participants | 0 | 1

7. Secondary Outcome: Corneal Re-epithelialization - Visit 2
Description: number of participants who had slit lamp photography which measured fluorescein staining size.
Time Frame: 16-day follow-up plus or minus 5 days
Measure: Number; unit: participants
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
participants | 1 | 2

8. Secondary Outcome: Corneal Re-epithelialization - Visit 3
Description: number of participants who had slit lamp photography which measured fluorescein staining size.
Time Frame: 30-day follow-up plus or minus 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

9. Secondary Outcome: Corneal Re-epithelialization - Visit 4
Description: number of participants who had slit lamp photography which measured fluorescein staining size.
Time Frame: 90-day follow-up plus or minus 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 1
Participants | 0 | 1

10. Secondary Outcome: Corneal Opacity Size - Visit 1
Description: number of participants who had anterior segment optical coherence tomography (ASOCT).
Time Frame: 5-day follow-up plus or minus 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
Participants | 1 | 1

11. Secondary Outcome: Corneal Opacity Size - Visit 3
Description: number of participants who had anterior segment optical coherence tomography (ASOCT).
Time Frame: 30-day follow-up plus or minus 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
Participants | 0 | 2

12. Secondary Outcome: Corneal Opacity Thinning-Visit 1
Description: number of participants who had anterior segment optical coherence tomography (ASOCT).
Time Frame: 5-day follow-up plus or minus 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
Participants | 1 | 1

13. Secondary Outcome: Corneal Opacity Thinning-Visit 3
Description: number of participants who had anterior segment optical coherence tomography (ASOCT).
Time Frame: 30-day follow-up plus or minus 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
Participants | 0 | 1

14. Secondary Outcome: Eye Pain- Visit 1
Description: Average pain rating across participants which was assessed subjectively using the Visual Analog Scale (VAS) ranging from 0 (none) to 10 (worst possible pain)
Time Frame: 5-day follow-up plus or minus 3 days
Population: All randomized subjects regardless of actual treatment, with data at the 5-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
score on a scale | 10 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 2.5 (1.5)

15. Secondary Outcome: Eye Pain- Visit 2
Description: as for outcome 14
Time Frame: 16-day follow-up plus or minus 5 days
Population: All randomized subjects regardless of actual treatment, with data at the 16-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
units on a scale | 1 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 1.7 (1.7)

16. Secondary Outcome: Eye Pain- Visit 3
Description: as for outcome 14
Time Frame: 30-day follow-up plus or minus 7 days
Population: All randomized subjects regardless of actual treatment, with data at the 30-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 2
units on a scale | 0 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 2 (2)

17. Secondary Outcome: Eye Pain- Visit 4
Description: as for outcome 14
Time Frame: 90-day follow-up plus or minus 10 days
Population: All randomized subjects regardless of actual treatment, with data at the 90-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 1
units on a scale | 2 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 0 (NA) — Standard deviation not available because only one participant was seen for visit 4. Participant not seen exited Prokera due to adverse event and was seen in clinic as part of standard of care only (Not study related).

18. Secondary Outcome: Eye Pain- Visit 5
Description: as for outcome 14
Time Frame: 180-day follow-up plus or minus 14 days
Population: All randomized subjects regardless of actual treatment, with data at the 180-day Follow-up Evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
Number analyzed (Participants) | 1 | 1
units on a scale | 0 (NA) — Standard deviation not available because only one participant is assigned conventional treatment. | 0 (NA) — Standard deviation not available because only one participant was seen for visit 4. Participant not seen excited Prokera due to adverse event and was seen in clinic as part of standard of care only (Not study related).

ADVERSE EVENTS:
Time Frame: 3 months
Description: The adverse event led to severe corneal melting resulting in emergency cornea transplants for 2/2 patients who received Prokera.
Arm/Group | Conventional Treatment | ProKera Plus® Treatment
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Treatment (N=1) | ProKera Plus® Treatment (N=2)
Corneal Melt (Eye disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This study was terminated early due to slow enrollment. There is not enough data collected for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT04850313/Prot_SAP_000.pdf